CLINICAL TRIAL: NCT05210140
Title: Utility of Plasma Drug Level Monitoring and CYP2C19 Genotyping in Dose Personalization of Escitalopram
Brief Title: Personalized Escitalopram Dosing in Patients With Depression
Acronym: PsyCise-E
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Collaborators: Clinical Centre of Serbia (Other); Institute of Mental Health, Serbia (Unknown); Military Medical Academy, Belgrade, Serbia (Other)
Responsible Party: Principal Investigator, Marin Jukic, Assistant Professor, PhD, University of Belgrade
Other Study IDs: 6066800-E
Record Dates: First submitted 2021-12-21; First posted 2022-01-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-01

CONDITIONS: Depressive Disorder, Major
Keywords: Escitalopram; Cytochrome p 450 cyp2c19; Precision medicine; Psychiatry; Pharmacogenetics; Serotonin Uptake Inhibitors
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two ml of plasma for the measurement of drug concentrations at visits at week 2, week 4 and week 8.
  Two ml of serum for biochemical analyses of liver and kidney function, cortisol levels, lipid status and glucose levels at visits at week 2, week 4 and week 8.
  "Buffy coat" taken from the 5 ml blood sample for DNA extraction and CYP2C19 genotyping, at any visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard dose: Patients are allocated to this group at visit V1 if 10 mg/day escitalopram treatment resulted in optimal escitalopram exposure (25-50 ng/ml) as measured at VK. These patients will continue their treatment with 10 mg/day during the V1-V2 period.
  Interventions: Drug: Escitalopram
- Adjusted dose: Patients are allocated to this group at visit V1 if 10 mg/day escitalopram dose resulted in to high (>50 ng/ml) or to low (<25 ng/ml) escitalopram exposure, as measured at VK. These patients will be treated with the adjusted escitalopram dose, different from 10 mg/day, during the V1-V2 period.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram, a selective serotonin reuptake inhibitor (SSRI), is commercially known as ELORYQA®, Elicea®, Escital®,PRAMES® or Lata® in Serbia. The recommended dose for Major depressive disorder is 10mg/day. Based on the individual response, dose can be adjusted and the maximum dose is 20 mg/day; 5 mg/day dose is also available. Escitalopram is also indicated for treatment of Obsessive-compulsive disorder, Generalized anxiety disorder, Social anxiety disorder (Social phobia) and Panic disorder (with or without agoraphobia) by Medicines and Medical Devices Agency of Serbia.
  In known CYP2C19 poor metabolizers, initial dose should be 5mg/day during first 2 weeks, and based on the individual response it can be increased up to maximum of 10 mg of escitalopram per day, according to the guidelines of Medicines and Medical Devices Agency of Serbia.
  Other Names: Lexapro; Citalex

SUMMARY:
The aims of this study are to:

1. Determine the proportion of participants who are underdosed or overdosed under recommended dosing regimen of escitalopram for the depression treatment (10 mg/day)
2. Determine and quantify clinical benefits of personalized escitalopram dosing regimen based on the escitalopram blood level monitoring
3. Retrospectively estimate whether the information on CYP2C19 genotype is useful in the prediction of escitalopram blood level.

DETAILED DESCRIPTION:
Escitalopram is an antidepressant extensively metabolized by the polymorphic CYP2C19 enzyme. Based on CYP2C19 genotype, patients can be classified either as:

* Normal metabolizers (Normal CYP2C19 enzyme capacity)
* Intermediate metabolizers (Decreased CYP2C19 enzyme capacity)
* Poor metabolizers (Absent CYP2C19 enzyme capacity)
* Ultra rapid metabolizers (Increased CYP2C19 enzyme capacity)

Adequate escitalopram exposure is needed to achieve optimal clinical response in the treatment of depression: too low drug plasma levels can lead to the lack of pharmacological effect, whereas too high drug plasma levels increases the incidence of adverse effects. There is evidence that patients with variant CYP2C19 genotypes have abnormal escitalopram exposure and could benefit from escitalopram dose personalization, but precise evidence-based protocol for personalized dosing of escitalopram has not been developed yet. This multicentric observational clinical trial is designed to collect crucial information for the development of such protocol that will be based on drug plasma level monitoring and/or CYP2C19 genotyping.

The course of the study will be as follows:

Initial Visit (V0):

Participant will be enrolled at this point if inclusion criteria are met. Escitalopram therapy will be initiated at the standard dose of 10 mg/day during next 2 weeks, or alternatively, started with 5 mg/day during first week and then increased to 10 mg/day during second week. General and socio-demographic information about the participant will be collected together with the baseline measurements: clinical questionnaires, anthropometric measurements, cardiology assessments, and the blood sample will be taken for biochemical analyses.

Mid-Visit (VK):

This visit takes place two weeks after the initial visit (V0) when escitalopram blood level is expected to reach the steady state. Blood sample will be taken from the participants at the end of the dose interval (before the morning dose) for the purpose of therapeutic drug monitoring. Plasma escitalopram levels will then be measured before the next visit and an independent clinician will allocate patients into one out of two cohorts based on whether or not escitalopram levels were optimal (25 - 50 ng/ml). If escitalopram levels were outside this interval, independent clinician will adjust the dose; escitalopram level lower than 5 ng/ml indicates noncompliance and results in dropout, level between 5 and 15 ng/ml results in dose increase to 20 mg/day, level between 15 and 25 ng/ml results in dose increase to 15 mg/day, level between 25 and 50 ng/ml results in treatment continuation with 10 mg/day, and level higher than 50 ng/ml results in dose decrease to 5 mg/day.

Visit 1 (V1):

Visit 1 takes place two weeks after VK and 4 weeks after the initiation of the escitalopram therapy. Without the knowledge of the attending clinician, independent clinician will adjust escitalopram doses accordingly. Attending clinician will then assess the participants using standardized questionnaires, participants will be anthropometrically and cardiologically examined, and blood samples will be taken for the purposes of therapeutic drug monitoring and biochemical analyses.

Visit 2 (V2):

Visit 2 is the final follow-up visit and it will be performed 4 weeks after the Visit 1 and 8 weeks after the escitalopram initiation. All participants will be assessed for psychometrical, anthropometrical and cardiological parameters, and blood samples will be taken again for the purposes of therapeutic drug monitoring and biochemical analysis.

If needed, additional participants, who are already on the stable escitalopram monotherapy, can be enrolled into study starting from VK. In this case, besides the blood sample for the therapeutic drug monitoring, all assessment usually done at initial visit (V0) will be performed during VK.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Major Depressive Disorder
* Starting monotherapy with escitalopram
* Signed written informed consent

Exclusion Criteria:

* Patient's requests to leave the study
* Patients who had taken escitalopram before
* Dementia
* Severe liver function impairment (abnormal AST/ALT ratio)
* Severe kidney function impairment (abnormal creatinine clearance)
* History of drug addiction (sporadic use is permitted)
* Suicide risk
* Patients who are taking strong CYP2C19 inhibitors
* Severe adverse drug reaction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population includes outpatients suffering from Major Depressive disorder who are previously untreated, and are seeking medical help for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depression severity score at week 8 | 8 Weeks
  Measured with clinician reported 21-item Hamilton rating scale for depression (HAM-D). Scale gives a score from 0 to 52 where higher score represents higher depression severity and worse outcome.
Adverse drug reaction severity score at week 8 | 8 Weeks
  Measured with clinician reported UKU (Udvalg for Kliniske Undersogelser) side effect rating scale. Scale gives summary score from 0 to 3 where higher scores correspond to the greater side-effects severity and worse outcome.

SECONDARY OUTCOMES:
Number of participants with escitalopram plasma concentrations outside the therapeutic window | at Week 2
  Therapeutic window is defined by escitalopram plasma concentrations of 25-50 ng/ml
Retrospectively determined regression formula for prediction of escitalopram plasma levels at Vk based on CYP2C19 metabolizer status | 8 Weeks
  CYP2C19 metabolizer status will be determined based on genotype as follows:
  Poor metabolizer: *2/*2, *2/*3, *3/*3
  Intermediate metabolizer: *1/*2, *1/*3
  Normal metabolizer: *1/*1
  Ultra-rapid metabolizer: *1/*17, *17/*17
  Several covariates will be considered: Body mass index, Creatinine clearance, AST/ALT ratio (Aspartate aminotransferase/Alanine aminotransferase)
Change from Baseline Depression severity score at week 4 | 4 Weeks
  Assessed with 21-item Hamilton rating scale for depression (HAM-D). Scale gives a score 0-52 where higher score is equivalent to the more severe depression and worse uotcome.
Adverse drug reaction severity score at week 4 | 4 Weeks
  Measured with clinician reported UKU (Udvalg for Kliniske Undersogelser) side effect rating scale. Scale gives summary score from 0 to 3 where higher scores correspond to the greater side-effects severity and worse outcome.

OTHER OUTCOMES:
Perception of stress score at baseline | Baseline
  Measured with self-reported Perceived stress scale (PSS). Scale gives scores from 0 to 40 where higher scores correspond to the higher severity of perceived stress and worse outcome.
Perception of stress score at week 4 | 4 Weeks
  Measured with self-reported Perceived stress scale (PSS). Scale gives scores from 0 to 40 where higher scores correspond to the higher severity of perceived stress and worse outcome.
Perception of stress score at week 8 | 8 Weeks
  Measured with self-reported Perceived stress scale (PSS). Scale gives scores from 0 to 40 where higher scores correspond to the higher severity of perceived stress and worse outcome.
Anxiety symptoms severity score at baseline | Baseline
  Measured with Hamilton anxiety rating scale (HAM-A). Scale gives scores from 0 to 56 where higher scores correspond to the higher severity of anxiety symptoms and worse outcome.
Anxiety symptoms severity score at week 4 | 4 weeks
  Measured with Hamilton anxiety rating scale (HAM-A). Scale gives scores from 0 to 56 where higher scores correspond to the higher severity of anxiety symptoms and worse outcome.
Anxiety symptoms severity score at week 8 | 8 Weeks
  Measured with Hamilton anxiety rating scale (HAM-A). Scale gives scores from 0 to 56 where higher scores correspond to the higher severity of anxiety symptoms and worse outcome.
Clinical Global Impression (CGI) Severity of illness score at baseilne | Baseline
  Measured with Clinical Global Impression scale for the severity of illness (CGI-S). Scale gives scores from 0 to 7 where higher scores correspond to the higher illness severity and worse outcome.
Clinical Global Impression (CGI) Severity of illness score at week 4 | 4 Weeks
  Measured with Clinical Global Impression scale for the severity of illness (CGI-S). Scale gives scores from 0 to 7 where higher scores correspond to the higher illness severity and worse outcome.
Clinical Global Impression (CGI) Severity of illness score at week 8 | 8 Weeks
  Measured with Clinical Global Impression scale for the severity of illness (CGI-S). Scale gives scores from 0 to 7 where higher scores correspond to the higher illness severity and worse outcome.
Clinical Global Impression (CGI) global improvement score at week 4 | 4 weeks
  Measured with Clinical Global Impression scale for the global improvement (CGI-I). Scale gives scores from 0 to 7 where higher scores correspond to the worse illness improvement and worse outcome.
Clinical Global Impression (CGI) global improvement score at week 8 | 8 weeks
  Measured with Clinical Global Impression scale for the global improvement (CGI-I). Scale gives scores from 0 to 7 where higher scores correspond to the worse illness improvement and worse outcome.
Clinical Global Impression (CGI) Efficacy index at week 4 | 4 weeks
  Measured with Clinical Global Impression scale - Efficacy index (CGI-E). Scale gives scores from 1 to 5 where higher scores correspond to the better outcome and beneficial drug efficacy/tolerability ratio.
Clinical Global Impression (CGI) Efficacy index at week 8 | 8 Weeks
  Measured with Clinical Global Impression scale - Efficacy index (CGI-E). Scale gives scores from 1 to 5 where higher scores correspond to the better outcome and beneficial drug efficacy/tolerability ratio.
Questionnaire of early childhood and recent traumatic experiences | Baseline
  Self-reported 13 item questionnaire by Pennebaker, J.W. & Susman, J.R. (1988)
QT interval at baseline | Baseline
  Determined on the electrocardiogram
QT interval at week 4 | 4 Weeks
  Determined on the electrocardiogram
QT interval at week 8 | 8 Weeks
  Determined on the electrocardiogram
Cortisol plasma levels at Baseline | Baseline
Cortisol plasma levels at week 4 | 4 Weeks
Cortisol plasma levels at week 8 | 8 Weeks
Employment status | Baseline
  Coded as follows:
  1. Unemployed,
  2. Employed; monthly incomes <40 000 RSD (~385$),
  3. Employed; monthly incomes 40 000-80 000 RSD (~385$-770$),
  4. Employed; monthly incomes >80 000 RSD (~770$).
Marital status | Baseline
  Coded as follows:
  1. Unmarried,
  2. Married,
  3. Divorced,
  4. Widowed
Education level | Baseline
  Coded as follows:
  1. Primary education (8 years),
  2. High school diploma (8+3 or 8+4 years),
  3. Associate's degree (8+4+2 or 8+4+3 years),
  4. Bachelor's degree (8+4+4 years) or higher

CONTACTS AND LOCATIONS:
Locations (3):
- Serbia (3):
  - Clinical Centre of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Institute of Mental Health, Belgrade

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared for all parameters relevant for two primary outcomes of this study.
  This will include, but is not limited to IPD data on: CYP2C19 metabolizer status and CYP2C19 genotype, HAM-D scores, UKU-scale scores and Escitalopram concentrations in the blood.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting from the time of publication of the main summary study results.
Access Criteria: IPD will be accessible to everyone.

REFERENCES:
- [Background] Pennebaker JW, Susman JR. Disclosure of traumas and psychosomatic processes. Soc Sci Med. 1988;26(3):327-32. doi: 10.1016/0277-9536(88)90397-8. PMID 3279521
- [Background] Jukic MM, Haslemo T, Molden E, Ingelman-Sundberg M. Impact of CYP2C19 Genotype on Escitalopram Exposure and Therapeutic Failure: A Retrospective Study Based on 2,087 Patients. Am J Psychiatry. 2018 May 1;175(5):463-470. doi: 10.1176/appi.ajp.2017.17050550. Epub 2018 Jan 12. PMID 29325448
- [Background] Milosavljevic F, Bukvic N, Pavlovic Z, Miljevic C, Pesic V, Molden E, Ingelman-Sundberg M, Leucht S, Jukic MM. Association of CYP2C19 and CYP2D6 Poor and Intermediate Metabolizer Status With Antidepressant and Antipsychotic Exposure: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 Mar 1;78(3):270-280. doi: 10.1001/jamapsychiatry.2020.3643. PMID 33237321

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05210140/Prot_SAP_000.pdf